CLINICAL TRIAL: NCT01649843
Title: Clinical Impact of Peroral Endoscopic Myotomy for Esophageal Achalasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Endoscopycenter-POEM
Record Dates: First submitted 2012-07-12; First posted 2012-07-25 (Estimated); Last update posted 2012-07-25 (Estimated); Status verified 2012-07

CONDITIONS: Esophageal Achalasia
Keywords: Peroral endoscopic myotomy; Esophageal Achalasia
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EA (Experimental): Patients were eligible for enrollment in the study if they had an Eckardt symptom score ≥ 4. The diagnosis of achalasia was made on the basis of the absence of peristalsis and on impaired relaxation of the LES on established methods (barium swallow, manometry, esophagogastroduodenoscopy (EGD)).
  Interventions: Procedure: POEM

INTERVENTIONS:
Procedure: POEM — Peroral endoscopic myotomy (POEM) has recently been described as a new minimally invasive endoscopic myotomy technique intending a permanent cure from primary achalasia in some centers.

SUMMARY:
Achalasia is a rare esophageal motility disorder, which is characterized clinically by symptoms of dysphagia, regurgitation, weight loss and chest pain. These symptoms are primarily caused by incomplete relaxation of a frequently hypertensive lower esophageal sphincter (LES) and to some extent by a lack of peristalsis in the tubular esophagus. Unfortunately, no therapy returns normal esophageal function. Treatment is therefore directed at lowering the LES pressure, with the aim of reducing the functional obstruction to bolus transit at this site. Current treatments can be endoscopic or surgical. Peroral endoscopic myotomy (POEM) has recently been described as a new minimally invasive endoscopic myotomy technique intending a permanent cure from primary achalasia in some centers. The investigators purpose was to further evaluate the efficacy and the feasibility of POEM for patients with achalasia in a prospective larger study.

DETAILED DESCRIPTION:
1. Patients were eligible for enrollment in the study if they had an Eckardt symptom score ≥ 4. The diagnosis of achalasia was made on the basis of the absence of peristalsis and on impaired relaxation of the LES on established methods (barium swallow, manometry, esophagogastroduodenoscopy (EGD)). Exclusion criteria were severe cardiopulmonary disease or other serious disease leading to unacceptable surgical risk, pseudoachalasia, and megaesophagus (diameter of > 7 cm).
2. All patients were scheduled for a follow-up visit at 1 month after POEM for EGD and manometry. Symptoms were assessed 1 month after treatment in the clinic and every 3 months thereafter via telephone questionnaires.
3. The primary outcome of the study was therapeutic success (a reduction in the Eckardt score to ≤3) at the follow-up assessment. The secondary outcomes included procedure-related adverse events, LES pressure on manometry pre- and post POEM, reflux symptoms and medication use before and after POEM, and procedure-related parameters such as procedure time, hospital stay, and myotomy length.

ELIGIBILITY:
Inclusion Criteria:

* with an Eckardt symptom score ≥ 4
* The diagnosis of achalasia was made on the basis of the absence of peristalsis and on impaired relaxation of the LES on established methods (barium swallow, manometry, esophagogastroduodenoscopy)
* Informed patient consent was obtained

Exclusion Criteria:

* Severe cardiopulmonary disease or other serious disease leading to unacceptable surgical risk
* Pseudoachalasia
* megaesophagus (diameter of > 7 cm)

Ages: 6 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Therapeutic success (a reduction in the Eckardt score to ≤3) | Symptoms were assessed 1 month after treatment in the clinic and every 3 months thereafter via telephone questionnaires during follow-up, an expected average of 2 years.

SECONDARY OUTCOMES:
Procedure-related adverse events | All patients were scheduled for a follow-up visit at 1 month after POEM for EGD.
Lower esophageal sphincter (LES) pressure on manometry | All patients were scheduled for a follow-up visit at 1 month after POEM for EGD and manometry
Reflux symptoms and medication use before and after POEM | Symptoms were assessed 1 month after treatment in the clinic and every 3 months thereafter via telephone questionnaires during follow-up, an expected average of 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hong Zhou, MD,PhD, Study Director — Endoscopy Center and Endoscopy Research Institute, Zhongshan Hospital, Fudan University, Shanghai, China
Locations (1):
- Endoscopy Center and Endoscopy Research Institute, Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Background] Eckardt AJ, Eckardt VF. Treatment and surveillance strategies in achalasia: an update. Nat Rev Gastroenterol Hepatol. 2011 Jun;8(6):311-9. doi: 10.1038/nrgastro.2011.68. Epub 2011 Apr 26. PMID 21522116
- [Result] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Result] von Renteln D, Inoue H, Minami H, Werner YB, Pace A, Kersten JF, Much CC, Schachschal G, Mann O, Keller J, Fuchs KH, Rosch T. Peroral endoscopic myotomy for the treatment of achalasia: a prospective single center study. Am J Gastroenterol. 2012 Mar;107(3):411-7. doi: 10.1038/ajg.2011.388. Epub 2011 Nov 8. PMID 22068665
- [Result] Ren Z, Zhong Y, Zhou P, Xu M, Cai M, Li L, Shi Q, Yao L. Perioperative management and treatment for complications during and after peroral endoscopic myotomy (POEM) for esophageal achalasia (EA) (data from 119 cases). Surg Endosc. 2012 Nov;26(11):3267-72. doi: 10.1007/s00464-012-2336-y. Epub 2012 May 19. PMID 22609984
- [Derived] Hu JW, Li QL, Zhou PH, Yao LQ, Xu MD, Zhang YQ, Zhong YS, Chen WF, Ma LL, Qin WZ, Cai MY. Peroral endoscopic myotomy for advanced achalasia with sigmoid-shaped esophagus: long-term outcomes from a prospective, single-center study. Surg Endosc. 2015 Sep;29(9):2841-50. doi: 10.1007/s00464-014-4013-9. Epub 2014 Dec 10. PMID 25492452